CLINICAL TRIAL: NCT03046043
Title: Ablation of Persistent Atrial Fibrillation Based on High Density Voltage Mapping and Complex Fractionated Atrial Electrogram
Brief Title: AF Ablation Based on High Density Voltage Mapping and CFAE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Principal Investigator, Hyoung-Seob Park, Associate Professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DSMCEP_PHS_002
Record Dates: First submitted 2017-02-03; First posted 2017-02-08 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2019-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-Voltage & CFAE guided ablation (Experimental): * Pulmonary isolation will be performed
  * Complex fractionated atrial electrogram(CFAE) and voltage mapping will be performed if atrial fibrillation the patient is still in atrial fibrillation after pulmonary vein isolation
  * CFAE and voltage mapping will be performed simultaneously using small electrode Pentaray® Catheter with CARTO®3 MEM version or CARTO®3 CONFIDENSE™
  * Automatic characterization of CFAE signals will be performed with an CARTO® CFAE software module.
  * CFAE areas within low voltage zone in the left atrium should be targeted first. If atrial fibrillation persist after left atrial ablation, target areas in the right atrium should be mapped and ablated. (Low-Voltage & CFAE guided ablation)
  Interventions: Procedure: pulmonary vein isolation; Procedure: Low-Voltage & CFAE guided ablation
- PV Isolation Only (Active Comparator): * Pulmonary vein isolation will be performed.
  * Electrical cardioversion to sinus rhythm will be performed if the patient is still in atrial fibrillation after pulmonary vein isolation.
  Interventions: Procedure: pulmonary vein isolation

INTERVENTIONS:
Procedure: pulmonary vein isolation — pulmonary vein isolation is conducted on the junction between the left atrium and pulmonary vein
Procedure: Low-Voltage & CFAE guided ablation — In CFAE guided ablation,. Within low voltage zone, CFAE areas defined by shortest SCI and high ICL are identified.-Areas with the shortest SCI and high ICL within low voltage areas should be targeted first, followed by longer SCI regions (up to 120ms). Radiofrequency energy is delivered at target sites for 30-60 sec until the local electrogram is completely eliminated.
  Arms: Low-Voltage & CFAE guided ablation

SUMMARY:
The purpose of this study is to evaluate the efficacy of additional ablation targeting complex fractionated atrial electrogram area within low voltage zone identified by high resolution mapping in patients with persistent atrial fibrillation.

DETAILED DESCRIPTION:
Fifty patients with persistent atrial fibrillation will be randomized a 1:1 ratio to each group. A test group includes those who undergoing ablation targeting low voltage areas which contains complex fractionated trial electrogram in addition to pulmonary vein isolation and a control group includes who undergoing pulmonary vein isolation only.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 20 years old and under 80 years old
2. Patients with non-valvular atrial fibrillation
3. Patients having atrial fibrillation even after receiving continued treatment with at least 1 antiarrhythmic drug for more than 6 weeks
4. Patients who can understand the information sheet and consent form on the need and procedure of catheter ablation and submitted them
5. Patients who are available of follow-up at least for more than three months after catheter ablation

Exclusion Criteria:

1. Patients unsuitable for catheter ablation because the size of left atrium is over 6.0 cm
2. Patients unsuitable for catheter ablation due to previous history of pulmonary surgery or structural heat disease.
3. Patients who cannot receive standard treatments such as anticoagulation therapy which need to be continuously performed prior to radiofrequency catheter ablation
4. Patients in the subject group vulnerable to clinical study
5. Patients who had undergone a prior catheter ablation for atrial fibrillation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Free from atrial arrhythmia at 12 months | 12 months
  Freedom from any atrial arrhythmia lasting longer than 30 seconds during 1 year follow-up after single ablation with or without the use of antiarrhythmic medications with the exclusion of the 3-month blanking period.

SECONDARY OUTCOMES:
Complication rate | 12 months
  Compare complication rate between two groups
Total procedure time, ablation time and fluoroscopy time | 12 months
  Compare total procedure time, ablation time and fluoroscopy time between two groups

CONTACTS AND LOCATIONS:
Overall Officials: Hyoung-Seob Park, MD, Principal Investigator — Keimyung University Dongsan Medical Center
Locations (1):
- Keimyung University Dongsan Medical Center, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided